CLINICAL TRIAL: NCT03782740
Title: Effect of Melatonin on Reduction of Pelvic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lena Marions, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mel PP
Record Dates: First submitted 2018-11-14; First posted 2018-12-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Dysmenorrhea; Endometriosis
MeSH Terms: conditions — Dysmenorrhea; Endometriosis | interventions — Melatonin; Sugars

STUDY DESIGN:
Intervention Model Description: Two parallel studies (dysmenorrhea and endometriosis) with 40 participants in each.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dysmenorrhea Melatonin 10 mg (Experimental): In the dysmenorrhea group: 2 capsules with 5 mg melatonin will be given in the evening for seven days consecutively during menstruation for two mentrual cycles. Compared with placebo.
  Interventions: Drug: Melatonin 10 mg; Drug: Placebo
- Endometriosis Melatonin 20 mg (Experimental): In the endometriosis group: 4 capsules with 5 mg melatonin will be given every evening during eight weeks. Compared with placebo.
  Interventions: Drug: Placebo; Drug: Melatonin 20 mg

INTERVENTIONS:
Drug: Melatonin 10 mg — Melatonin capsule
  Other Names: N-acetyl-5-methoxy tryptamine
  Arms: Dysmenorrhea Melatonin 10 mg
Drug: Placebo — Sugar pill manufactured to mimic Melatonin capsule
  Other Names: Sugar pill
Drug: Melatonin 20 mg — Melatonin capsule
  Other Names: N-acetyl-5-methoxy tryptamine
  Arms: Endometriosis Melatonin 20 mg

SUMMARY:
In two double blinded randomized controlled trials (RCT) we will study the effect of pain reduction of melatonin vs placebo in women with severe dysmenorrhea and women with endometriosis.The aim is to find an effective method for pelvic pain caused by dysmenorrhea and endometriosis.The primary outcome is reduction of pain in patients with dysmenorrhea and endometriosis respectively when treated with melatonin vs placebo. Secondary outcomes include the effect on daily life, quality of life and cognition. Sleep will also be assessed to evaluate its potential relation to quality of life and cognition.

DETAILED DESCRIPTION:
Two substudies will be performed. Forty women with severe dysmenorrhea will be randomized to treatment with 10 mg melatonin daily or placebo during the menstruation for 2 menstrual cycles. Another 40 women with endometriosis will be randomized to treatment with 20 mg or placebo daily during 8 weeks. Participants will report drug intake, bleeding details (duration and amount) and pain as well as possible side effects. They will also perform a test for sleep quality and cognition before and after completion of the study.

See protocol for more details

ELIGIBILITY:
Dysmenorrhea group

Inclusion Criteria:

* Regular menstrual cycles,
* Severe dysmenorrhea (NRS>6)
* Speaks and understands Swedish
* If other medication, those should be un-altered for the last 3 months

Exclusion Criteria:

* Smoker
* Prior or ongoing liver or kidney disease
* Endometriosis
* Pregnancy

Endometriosis group:

Criteria for inclusion:

* Endometriosis (endometriomas or diagnosis by laparoscopy)
* Moderate to severe pain (NRS >/= 4)
* Good general health
* Understands and speaks Swedish
* If any other treatment, unchanged regimen for the last 3 months
* Signed informed consent

Criteria for exclusion:

* Prior or ongoing disease in kidney or liver
* Use of opioid analgesics
* Smoker
* Pregnant

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 12 weeks
  Self reported pain intensity daily, Numeric Rating Scale (NRS) 0-10 (0=no pain, 10 = worst possible pain)

SECONDARY OUTCOMES:
Use of analgesics | 12 weeks
  Self reported daily quantification of intake of analgesics reported online
Quality of sleep | 12 weeks
  Insomnia Severity index questionnaire will be administered during observational cycle and once during the second treatment cycle. 0 to 28 Points, 0-7 Points signifies no Clinical significant sleeping dificulties, 22-28 Points signifies Clinical insomnia)
Cognition | 12 weeks
  Dysmenorrhea group: Online test (CANTAB) performed on day 1-4 in the menstrual cycle in the observational cycle and in the second treatment cycle.
Catastrophic thinking | 12 weeks
  Endometriosis group: Pain Catastrophizing Scale questionnaire will be administered during observational cycle and once during the second treatment cycle. 0-52 Points, higher points indicate higher tendency to catastrophize.
General well being | 12 weeks
  Endometriosis group: Quality of life assessment with Endometriosis Health Profile (EHP-30) will be administered during observational cycle and once during the second treatment cycle. Score 0-100 Points, where 0 is best health status and 100 is worst health status.
Acceptance of Melatonin | 12 weeks
  Assessment at the end of study
Side effects of Melatonin | 12 weeks
  Online self reporting, daily

CONTACTS AND LOCATIONS:
Locations (1):
- Södersjukhuset, Stockholm, Sweden

REFERENCES:
- [Derived] Soderman L, Bottiger Y, Edlund M, Jarnbert-Pettersson H, Marions L. Adjuvant use of melatonin for pain management in endometriosis-associated pelvic pain-A randomized double-blinded, placebo-controlled trial. PLoS One. 2023 Jun 2;18(6):e0286182. doi: 10.1371/journal.pone.0286182. eCollection 2023. PMID 37267394
- [Derived] Soderman L, Edlund M, Bottiger Y, Marions L. Adjuvant use of melatonin for pain management in dysmenorrhea - a randomized double-blinded, placebo-controlled trial. Eur J Clin Pharmacol. 2022 Feb;78(2):191-196. doi: 10.1007/s00228-021-03234-6. Epub 2021 Oct 20. PMID 34668986